CLINICAL TRIAL: NCT01207596
Title: Evaluating the Efficacy and Safety of Extended Release Hydromorphone (Exalgo) in Patients With Neuropathic Pain: An Open Label Study
Brief Title: Evaluating the Efficacy and Safety of Extended Release Hydromorphone (Exalgo) in Patients With Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Srinivas Nalamachu, MD, International Clinical Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-NP2010
Record Dates: First submitted 2010-09-20; First posted 2010-09-23 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Neuropathic Pain
Keywords: Pain; Neuropathy; Neuropathic Pain; Hydromorphone
MeSH Terms: conditions — Neuralgia; Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydromorphone (Active Comparator)
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Oral hydromorphone extended release, once daily
  Other Names: EXALGO (R)

SUMMARY:
The purpose of this study is to find out if Exalgo (r) is beneficial for the patients with neuropathic pain.

DETAILED DESCRIPTION:
Neuropathic pain state is usually refractory to most analgesic regimens and requires polypharmacy for symptomatic relief. Current treatment options for neuropathic pain include both oral and topical medications. Most commonly prescribed oral treatments include antidepressants (eg, amitriptyline, desipramine, and duloxetine), antiepileptics (eg, gabapentin, pregabalin), and opiates such as tramadol and morphine. Current topical treatments include the lidocaine patch and the capsaicin patch. Many patients have inadequate pain relief in spite of these treatment options.

Currently, there are no treatments available for treatment of neuropathy itself other than treating the underlying cause and addressing the symptomatic relief for pain. Current drug therapies for neuropathic pain provide inadequate pain relief and undesirable side effects including sedation and cognitive dysfunction. It is not uncommon to use a combination of agents for the treatment of neuropathic pain to minimize the side effects. Although treating the mild to moderate pain may be relatively easy, it is very challenging for severe neuropathic pain. Although the use of opiates for neuropathic pain is well accepted, it remains controversial because of the potential for abuse and diversion.

ELIGIBILITY:
Inclusion Criteria:

1. individuals with chronic pain of more than 6 months duration
2. pain is determined to be secondary to a documented neuropathy
3. patients who are tolerant of opiates (60 mg of morphine or equivalent for at least one week)
4. male or female patients aged 18-75 yrs and have signed a written informed consent form and privacy statement
5. female patients of child-bearing potential must be using an acceptable form of birth control

Exclusion Criteria:

1. pregnant or lactating women
2. allergy to morphine or its derivatives
3. history of alcohol or substance abuse in the last 3 yrs
4. participation in any other clinical trial in the last 30 days
5. uncontrolled pain
6. patient who is deemed to be medically unstable by principal investigator
7. history of severe lung disease or asthma that is deemed medically significant by principal investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research Institute
Locations (1):
- International Clinical Research Institute, Leawood, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone: Received once-daily OROS hydromorphone ER, individually titrated, available in 8, 12, and 16-mg tablet strengths
Period: Overall Study
Arm/Group | Hydromorphone
Started | 30
Completed | 21
Not Completed | 9
Not completed — Physician Decision | 4
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hydromorphone
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Pain Over the Last 24 Hrs on the Brief Pain Inventory (BPI) Scale
Description: The primary efficacy measure was the change from baseline to end of study on question #5 ("average pain") of the Brief Pain Inventory (BPI): "Please rate your pain by marking the box beside the number that best describes your pain on the average," where 0 = no pain and 10 = pain as bad as you can imagine.
Time Frame: Baseline visit to Week 12 or last visit
Population: LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
units on a scale | -1.2 (0.55)

2. Secondary Outcome: Change From Baseline in the Average Pain Over the Last 24 Hrs on the Brief Pain Inventory (BPI) Scale Question #3: the Number That Best Describes Your Pain at Its Worst in the Last 24 Hours
Description: Change from baseline to end of study on question #3 ("worst pain") of the Brief Pain Inventory (BPI): "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the last 24 hours," where 0 = no pain and 10 = pain as bad as you can imagine.
Time Frame: Baseline visit to Week 12 or last visit
Population: LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
units on a scale | -1.8 (0.61)

3. Secondary Outcome: Change From Baseline in the Average Pain Over the Last 24 Hrs on the Brief Pain Inventory (BPI) Scale Question #4: the Number That Best Describes Your Pain at Its Least in the Last 24 Hours
Description: Change from baseline to end of study on question #4 ("least pain") of the Brief Pain Inventory (BPI): "Please rate your pain by marking the box beside the number that best describes your pain at its least in the last 24 hours," where 0 = no pain and 10 = pain as bad as you can imagine.
Time Frame: Baseline visit to Week 12 or last visit
Population: LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
units on a scale | -0.9 (0.57)

4. Secondary Outcome: Change From Baseline in the Average Pain Over the Last 24 Hrs on the Brief Pain Inventory (BPI) Scale Question #6: the Number That Tells How Much Pain You Have Right Now
Description: Change from baseline to end of study on question #4 ("current pain") of the Brief Pain Inventory (BPI): "Please rate your pain by marking the box beside the number that tells how much pain you have right now," where 0 = no pain and 10 = pain as bad as you can imagine.
Time Frame: Baseline visit to Week 12 or last visit
Population: LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
units on a scale | -1.3 (0.59)

5. Secondary Outcome: Sleep Quality Assessment (SQA)
Description: Sleep Quality Assessment (SQA) scale, asking patients to assess the degree that pain has interfered with their sleep in the last 24 hours (where 0 = does not interfere and 10 = completely interferes)
Time Frame: Baseline visit to Week 12 or last visit
Population: LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
units on a scale | -1.7 (0.60)

6. Secondary Outcome: Pain Quality Assessment Scale (PQAS)
Description: The PQAS is a 20-item scale that quantifies the quality and intensity of neuropathic and non-neuropathic pain; scores range from 1 to 200, with higher scores indicating more severe pain
Time Frame: Baseline visit to 12 weeks visit
Population: LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
units on a scale | -24.8 (7.9)

7. Secondary Outcome: Global Assessment of Treatment Satisfaction
Description: Patients were asked to rate their global assessment of treatment satisfaction, ranging from "very dissatisfied" to "very satisfied". Adverse events were monitored throughout the study
Time Frame: Baseline visit to Week 12 or last visit
Population: LOCF
Measure: Number; unit: percentage of patients
Arm/Group | Hydromorphone
Number analyzed (Participants) | 26
percentage of patients
  Very satisfied | 38.5
  Satisfied | 42.3
  Dissatisfied | 15.4
  Very dissatisfied | 3.8

ADVERSE EVENTS:
Arm/Group | Hydromorphone
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 11/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone (N=30)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (4)
Flu (Gastrointestinal disorders) | 3 (3)
Increased pain (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No